CLINICAL TRIAL: NCT00879463
Title: The Impact of Brain Tissue Oxygen Saturation Monitoring in Reducing the Use of Red Blood Cells in Cardiac Surgery
Brief Title: Brain Tissue Oxygen Saturation and Blood Transfusion in Cardiac Surgery
Acronym: INVOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, STAVROULA GEORGOPOULOU, MD, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UH 1969 TT
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Blood Transfusion; Cardiac Surgery
Keywords: Blood transfusion in cardiac operations under CPB; Infrared spectrophotoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP A (Active Comparator): Brain tissue oxygen saturation monitoring
  Interventions: Procedure: Brain tissue oxygen saturation monitoring
- GROUP B (Active Comparator): CONTROL GROUP
  Interventions: Procedure: Transfusion according to the anesthesiologist's judgement

INTERVENTIONS:
Procedure: Brain tissue oxygen saturation monitoring — Brain tissue oxygen saturation monitoring with infrared spectrophotoscopy
  Arms: GROUP A
Procedure: Transfusion according to the anesthesiologist's judgement — Transfusion if hemoglobin is between 5.5-7 mg/dl
  Arms: GROUP B

SUMMARY:
In cardiac operations under cardiopulmonary bypass(CPB), monitoring of brain tissue oxygen saturation with infrared spectrophotoscopy leads to a reduction of the number of packed red cell(PRC) transfusions during the period of extracorporeal circulation.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether the use of brain tissue oxygen saturation monitoring will lead to a reduction of the intra-operative use of packed red cell units.

Patients randomly allocated to groups A and B. In group A INVOS monitoring available. In group B, no access to INVOS for the attending anesthesiologist. An "observer" anesthesiologist has access to INVOS and provides information if it is considered necessary.

For BOTH GROUPS:

During CBP and before aortic unclamping, PRC not to be given if hemoglobin is >7g/dl. For values less than 5.5g/dl, one unit of PRC is transfused and the patient is reevaluated. After weaning from CPB and retransfusion of the salvaged shed blood, transfusion when hemoglobin is <8g/dl. During ICU stay, transfusion when hemoglobin is <8g/dl. Between 8-10g/dl evaluation for transfusion in a multimodal manner.

For GROUP A:

As above and during CBP and before aortic unclamping, if hemoglobin is between 5.5-7g/dl, transfusion when INVOS is less than 60%.

For GROUP B:

As above and during CBP and before aortic unclamping, if hemoglobin is between 5.5-7g/dl, decision for transfusion is taken by the attending anesthesiologist (judgment).

ELIGIBILITY:
Inclusion Criteria:

* Cardiac operations under cardiopulmonary bypass, consequently (including coronary-aortic bypass graft), valve replacement, surgery of the ascending aorta, combined procedures, redo-operations)

Exclusion Criteria:

* Cardiac operations without the aid of extracorporeal circulation (ex. "off-pump" techniques)
* Emergency operations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The number of packed red cell units transfused intra-operatively | one year

SECONDARY OUTCOMES:
The INVOS values electronically and continuously | one year
The volume of any kind of intravenous fluids administered to the patient | one year
The volume of urine output from the initiation to termination of CPB and to the end | one year
The hematocrit values at certain timeframes | one year

CONTACTS AND LOCATIONS:
Overall Officials: STAVROULA GEORGOPOULOU, M.D., Principal Investigator — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; GEORGE VRETZAKIS, M.D. PhD, Study Director — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; KONSTANTINOS STAMOULIS, MD, Study Chair — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece; ATHINA KLEITSAKI, MD, Study Chair — Cardiac Anesthesia Unit, Department of Anesthesiology, University Hospital of Larissa, Greece
Locations (1):
- Larissa University Hospital, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Goodnough LT, Shander A. Evolution in alternatives to blood transfusion. Hematol J. 2003;4(2):87-91. doi: 10.1038/sj.thj.6200237. No abstract available. PMID 12750725
- [Background] Tinmouth A, Macdougall L, Fergusson D, Amin M, Graham ID, Hebert PC, Wilson K. Reducing the amount of blood transfused: a systematic review of behavioral interventions to change physicians' transfusion practices. Arch Intern Med. 2005 Apr 25;165(8):845-52. doi: 10.1001/archinte.165.8.845. PMID 15851633
- [Derived] Vretzakis G, Georgopoulou S, Stamoulis K, Tassoudis V, Mikroulis D, Giannoukas A, Tsilimingas N, Karanikolas M. Monitoring of brain oxygen saturation (INVOS) in a protocol to direct blood transfusions during cardiac surgery: a prospective randomized clinical trial. J Cardiothorac Surg. 2013 Jun 7;8:145. doi: 10.1186/1749-8090-8-145. PMID 23758929